CLINICAL TRIAL: NCT04400968
Title: A Randomised Clinical Trial of the Effects of Kinesiotaping vs.Auricular Therapy in Women With Primary Dysmenorrhoea.
Brief Title: Effects of Kinesiotaping vs.Auricular Therapy in Primary Dysmenorrhoea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, PHD, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58/2017
Record Dates: First submitted 2020-05-09; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Primary Dysmenorrhoea
Keywords: auricular therapy; kinesio tape
MeSH Terms: interventions — Acupuncture, Ear; Auriculotherapy; Athletic Tape

STUDY DESIGN:
Intervention Model Description: Double-blind randomized clinical controlled trial. Participants were randomized to a auricular therapy group, an auricular therapy placebo group, a kinesio tape group, a kinesio tape placebo group and a control group for a 11 month study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants in the different intervention groups received real and placebo auricular therapy and kinesio tape treatment.
  The kinesio tape placebo group had the application of three elastic bandages that were shorter than the used in the kinesio tape group. In addition, the tape was adhered with no tension and not place in the treatment area. The auricular therapy placebo group had adhesive tapes without seeds displaced from the treatment points.
  The outcome assessor was independent to the study and was not aware of the treatments applied or the objective of the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Auricular therapy group (Experimental): The auricular therapy group received an intervention based on the bilateral application of 7 adhesive tapes with vaccaria seeds. The points were located with a retractable 250 gr. pressure palpator (Sedatelec®). An experienced health professional trained on acupuncture techniques applied the vaccaria seeds.
  Interventions: Procedure: Auricular therapy
- Auricular therapy Placebo group (Sham Comparator): The auricular therapy placebo group had adhesive tapes without seeds displaced from the treatment points.
  Interventions: Procedure: Auricular therapy Placebo group
- Kinesio tape group (Experimental): The kinesio tape group received an intervention that consisted on the standard application of three elastic bandages. An experienced kinesio tape certified physical therapist applied the taping.
  Interventions: Procedure: kinesio tape
- kinesio tape Placebo group (Sham Comparator): The kinesio tape placebo group had the application of three elastic bandages that were shorter than the used in the kinesio tape group. In addition, the tape was adhered with no tension and not place in the treatment area.
  Interventions: Procedure: kinesio tape Placebo group
- Control group (No Intervention): The control group did not receive any treatment. The participants continued with their routine medical treatment. However, the controls completed all the questionnaires to collect the information regarding their symptoms in order to observe their progress with no intervention.

INTERVENTIONS:
Procedure: Auricular therapy — The auricular therapy points were selected following the protocol for dysmenorrhoea described by Oleson (Oleson, 2008). These points were (the name of the European cartography is specified by the name of the point): Shenmen [FT2], uterus [FT5], sympathetic [HI4], kidney [CS6], heart [CI4], endocrine [IT2] and thalamus [PC2].
  Other Names: Auricular acupuncture; ear therapy; auriculotherapy
  Arms: Auricular therapy group
Procedure: kinesio tape — Before the tape application, the skin surface was removed of hair when needed and cleansed. The tapes were applied at 25% of tension and were placed horizontally covering the area between the antero-superior iliac spines and the postero-superior iliac spines and vertically from the navel to the symphysis pubis. All bandages were adhered to the skin with a technique type I with a space augmentation. The centre of the tape was removed and applied at 25% of tension. Afterwards, the rest of the protector were removed and the laterals anchors of the tape were adhered with no tension. The participant maintained a slight extension of the trunk while the tape was applied on the anterior aspect of the truck and a slight flexion while the tape was applied in the posterior aspect of the trunk.
  Other Names: medical taping concept; neuromuscular taping
  Arms: Kinesio tape group
Procedure: Auricular therapy Placebo group — Sham auricular therapy
  Arms: Auricular therapy Placebo group
Procedure: kinesio tape Placebo group — Sham kinesio tape
  Arms: kinesio tape Placebo group

SUMMARY:
This study analyse the effectiveness of auricular therapy vs. kinesio tape treatment for pain management of women with primary dysmenorrhoea.

DETAILED DESCRIPTION:
Pharmacological treatments are not effective for all women and therefore, the objective of this study was to assess and compare the effectiveness of kinesio tape and auricular therapy to decrease pain and drug intake in women with primary dysmenorrhoea.

A randomized controlled trial was conducted. 114 university women from 18 to 30 years old were randomized to 5 groups: control, kinesio tape, placebo kinesio tape, auricular therapy and placebo auricular therapy. The study was carried out during 4 menstrual cycles of pre-treatment phase, 4 menstrual cycles of treatment phase and two follow up phases (first and third cycle after the treatments were completed). During the treatment phase, the techniques were applied during 72h in each cycle.

The primary outcome measures were: Mean pain intensity of the 3 first days of bleeding, maximum pain intensity, number of painful days and dose of drug intake measured with the Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 30 years old affected by primary dysmenorrhoea grade 2 and 3 of Andersch y Milsom classification (Andersch y Milsom, 1982), to have attended gynaecologist consultation for a general revision in the last 2 years, to have menstrual pain, to have regular menstrual cycles of 21 to 38 days, to not have an intrauterine/inter-uterine) device or to be on oral contraceptive treatment.

Exclusion Criteria:

* To have been diagnosed with a condition that could influence menstrual pain perception, to know or have been previously treated with the techniques used in the interventions and pregnancy.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with Primary dysmenorrhoea , a pathology that only affects women
Enrollment: 160 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Changes from the Mean pain intensity | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Mean pain intensity of the 3 first days of menstruation measured with the Visual Analogue Scale. Scores range from 0 to 10 where where 0 means no pain and 10 means maximum and excruciating pain.
Changes from the Maximum pain intensity | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Maximum pain intensity during menstruation measured with the Visual Analogue Scale. Scores range from 0 to 10 where where 0 means no pain and 10 means maximum and excruciating pain.
Changes from number of painful days | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Count of number of days when the participant experienced pain during the menstruation. A lower number of painful days indicate an improvement
Changes from the dosage of drug intake | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Register of dosage and grug intake of each participant to relief pain during the menstruation. A lower dose of drug intake indicate an improvement.

SECONDARY OUTCOMES:
Changes from the Length of the menstrual cycle | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Count of days that the menstrual cycle lasted for.
Changes from the Length of menstruation | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Count of days that menstruation lasted for.
Changes from theType of drug | Measured at the end of the menstruation of 4 cycles (28 days) during the pre-treatment and the treatment phase (total of 8 measurements) and at the end of the menstruation of the 9th and 11th cycle (Follow up)
  Record of type of medication used by the participants during the menstruation for pain relief.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No